CLINICAL TRIAL: NCT05973578
Title: Cardiac RadiothErapy for VEntricular Tachycardia
Acronym: CREVET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s66934
Record Dates: First submitted 2023-05-02; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-05

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic body radiotherapy (Other): Patients will be treated with a stereotactic body radiotherapy technique as a single fraction treatment up to a dose of 25 Gy delivered to the VT substrate
  Interventions: Radiation: Stereotactic radiotherapy

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — Single-session high dose stereotactic radiotherapy

SUMMARY:
Objective: To explore in our center the feasibility and safety of a SBRT treatment method for VT.

Study population: Patients with ventricular tachycardia that are refractory to dose-escalated antiarrhythmic drugs and where catheter ablation has either already been performed or is deemed to be unsuccessful or associated with high risks.

Intervention: Patients will be treated with a stereotactic body radiotherapy technique as a single fraction treatment up to a dose of 25 Gy delivered to the VT substrate defined by electrophysiological mapping.

Main study endpoints: The primary aim is to explore the feasibility and safety of a SBRT treatment method for refractory VT. Secondary endpoints include an assessment of the efficacy of the treatment, quality of life, late toxicity and overall survival.

Patients will have to fill in a quality-of-life questionnaire before and after the radiotherapy treatment. The risk associated with this trial is an increase in toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years
* Presence of a structural heart disease and an implantable cardioverter defibrillator (ICD)
* Documented sustained monomorphic VT that requires ICD intervention (e.g., shock or anti-tachycardia stimulation)
* The VT is inducible by ICD via non-invasive programmed stimulation (NIPS) or during electrophysiology measurement
* Patient must have failed or become intolerant to at least one antiarrhythmic medication
* Patient must have failed at least one invasive catheter ablation procedure, or have a contraindication to a catheter ablation procedure, or have VT thought to arise from a protected location
* Ability to give a written informed consent and willingness to return for follow-up

Exclusion Criteria:

* Pregnancy or breastfeeding
* Lack of evidence of a myocardial scar triggering the VT
* Polymorphic VT or ventricular fibrillation (VF) as a clinical heart rhythm
* Advanced symptomatic heart failure defined as NYHA Class IV heart failure
* Previous radiotherapy with cardiac involvement
* Life expectancy < 6 months, in the absence of VT, as best based on clinical judgment by the treating and enrolling physicians
* Any condition that is deemed a contraindication in the judgment of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of SBRT | From date of inclusion up to 1 year
  Successful irradiation process (collaboration with cardiologist and radiologist), measured by the end-to-end delivery of SBRT to at least 1 patient
Safety of SBRT | From radiotherapy up to 1 year
  Measurement of acute and late toxicity assessed using the CTCAE v5.0

SECONDARY OUTCOMES:
Efficacy of SBRT | From inclusion up to 1 year
  Changes in the use of antiarrhythmic medication, reduction in VT burden
Health related quality-of-life | From inclusion up to 1 year
  Measurement of the quality of life using the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No